CLINICAL TRIAL: NCT06451198
Title: IndObufen Versus asPirin After Coronary Drug-eluting Stent implantaTION in Elderly Patients With Acute Coronary Syndrome
Acronym: OPTION2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-187
Record Dates: First submitted 2024-06-03; First posted 2024-06-11 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — indobufen; Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- indobufen plus ticagrelor (Experimental): Patients meeting the criteria are randomized before discharge from the hospital and given indobufen 100 mg bid and ticagrelor 90mg bid the second day after randomization. The administration shall last 12 months.
  Interventions: Drug: Indobufen; Drug: Ticagrelor
- aspirin plus ticagrelor (Active Comparator): Patients meeting the criteria are randomized before discharge from the hospital and continued aspirin 100 mg qd and ticagrelor 90mg bid. The administration shall last 12 months.
  Interventions: Drug: Aspirin; Drug: Ticagrelor

INTERVENTIONS:
Drug: Indobufen — Patients meeting the criteria are randomized before discharge from the hospital and given indobufen 100mg bid and ticagrelor 90mg bid the second day after randomization. The administration shall last 12 months.
  Arms: indobufen plus ticagrelor
Drug: Aspirin — Patients meeting the criteria are randomized before discharge from the hospital and continued aspirin 100 mg qd and ticagrelor 90mg bid. The administration shall last 12 months.
  Arms: aspirin plus ticagrelor
Drug: Ticagrelor — All the patients meeting the criteria and enrolled in the study are given ticagrelor 90mg bid for 12 months.

SUMMARY:
The OPTION2 trial (randomized controlled trial of IndObufen versus asPirin after coronary drug-eluting stent implantaTION in elderly patients with acute coronary syndrome) was designed to compare the 1-year clinical efficacy and safety of indobufen-based dual antiplatelet therapy (DAPT) (indobufen 100mg bid plus ticagrelor 90mg bid) or conventional DAPT (aspirin 100mg qd plus ticagrelor 90mg bid) in acute coronary syndrome (ACS) patients aged over 70 years old undergoing coronary drug-eluting stent (DES) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 70 years old
* Diagnosed with acute coronary syndrome (unstable angina/ non-ST elevation myocardial infarction/ ST elevation myocardial infarction)
* Treated with at least 1 DES implanted in the coronary lesion
* Receiving dual antiplatelet therapy (aspirin plus ticagrelor)
* Agree to attend the trial

Exclusion Criteria:

* Elective surgical procedure planned within 12 months
* Life expectancy ≤1 year
* Known allergy or intolerance to aspirin, ticagrelor or nonsteroidal anti-inflammatory drugs (NSAIDs)
* History of cerebral hemorrhage
* History of stroke in six months
* Active bleeding
* Known relevant hematological deviations
* Known, clinically important thrombocytopenia (i.e., <100*10^9/L) or anemia (i.e., <90g/L)
* Active cancer
* Concomitant use of oral anticoagulants
* Active participation in another clinical study
* Other situations in which the investigator considers unsuitable to attend the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2846 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
net adverse clinical events (NACEs) | 1-year
  including ischemic and bleeding events, i.e., a composite of cardiovascular (CV) death, nonfatal myocardial infarction (MI), ischemic stroke, definite or probable stent thrombosis (ST), or Bleeding Academic Research Consortium (BARC) criteria type 2, 3 or 5 bleeding

SECONDARY OUTCOMES:
a composite of CV death, nonfatal MI, ischemic stroke, definite or probable ST | 1-year
  ischemic events
BARC criteria type 2, 3 or 5 bleeding events | 1-year
  bleeding events
a composite endpoint of CV death, nonfatal MI, ischemic stroke, definite or probable ST, or BARC criteria type 3 or 5 bleeding | 1-year
  key composite endpoint
all-cause mortality | 1-year
  death from any cause

IPD SHARING:
Plan to Share IPD: No